CLINICAL TRIAL: NCT04007848
Title: Cobimetinib for BRAF-wild-type or Mutated Histiocytoses : a Randomized, Placebo-controlled, Double Blind Study" COBRAH Study
Brief Title: Cobimetinib for BRAF-wild-type or Mutated Histiocytoses
Acronym: COBRAH
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P170932J - 2018-00222-23
Record Dates: First submitted 2019-06-18; First posted 2019-07-05 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2024-12

CONDITIONS: Disease or R Group Histiocytoses
MeSH Terms: conditions — Disease | interventions — cobimetinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cobimetinib (Experimental): Experimental group : 36 histiocytoses's patients without or with BRAF V600E will be randomised in cobimetinib group
  Interventions: Drug: Cobimetinib
- Placebo (Placebo Comparator): Control group : 18 histiocytoses's patients without or with BRAF V600E will be randomised in the placebo group
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Cobimetinib — Cobimetinib will be given at the dose of 40 milligrams once a day (21 days/28). Cobimetinib is available as 20 milligrams film-coated tablets
  Other Names: COTELLIC
  Arms: Cobimetinib
Drug: Placebo oral tablet — Placebo will be given at the dose of 40 milligrams once a day (21 days/28). Placebo is available as 20 milligrams film-coated tablets
  Other Names: PLACEBO
  Arms: Placebo

SUMMARY:
COBRAH is a randomized double-blind 2-steps controlled superiority trial, with 2 parallel groups.

Patients will be randomly assigned in a 2:1 ratio to receive Cobimetinib orally or placebo during the first 12-weeks step, allowing the determination of the primary criteria.

DETAILED DESCRIPTION:
Histiocytoses are rare multisystemic disorders characterized by accumulation of histiocytes in various organs. Virtually all the patients have a somatic mutation in the RAS-RAF-MEK-ERK pathway. BRAF inhibitors are efficacious to treat BRAF-mutated patients but one third of the patients are BRAF-wild type. For these patients, preliminary data have shown an efficacy of the MEK inhibitor cobimetinib. This trial aims to evaluate the efficacy of cobimetinib for treating BRAF-wild type or mutated patients with L or R group histiocytoses.

The primary objective of the COBRAH trial is to demonstrate that the rate of objective metabolic response (complete or partial) according to PERCIST criteria is higher under Cobimetinib versus placebo.

The objective metabolic response according to PERCIST criteria (Haroche, et al. 2015) is defined by the Positron Emission Tomography (PET) response and will be used to evaluate the overall therapeutic response at month 3 (Week 12).

For PERCIST criteria, a quantitative analysis of uptake will be performed using the standard uptake value (SUV). Fitting regions of interest covering pathologic uptake will be used to define target lesions. PERCIST will be used to classify the patients as complete metabolic response, partial metabolic response (reduction of a minimum of 30% in target lesions), stable metabolic disease or progressive metabolic disease.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients should be at least 18 years of age,
* Have a histologically confirmed L or R group histiocytoses without BRAFV600E mutation detected with the use of a real-time polymerase chain reaction or with BRAFV600E mutation AND a contra-indication to BRAF inhibitors
* Have a measurable disease according to the PERCIST criteria with presence of at least one severe organ involvement (heart, vascular, central nervous system) OR a multisystemic disease with ≥3 organ involvement AND failure of a first-line treatment or contra-indication to these treatments,
* Accepting effective contraception during treatment duration (men and women childbearing potential) and 3 months after.
* Signed informed consent

Exclusion Criteria:

* Patients with severe hepatic, renal and cardiac outcomes
* Patients with myopathies at baseline
* Patients with retinal detachment at baseline
* Patients with inherited disorders of galactose intolerance, Lapp lactase deficiency or glucose-galactose malabsorption
* Patients with high bleeding risk.
* Allergies to iodized contrast media
* Simultaneous participation in another medical research
* Pregnancy or breast-feeding.
* No affiliation to the French Health Care System "sécurité sociale" OR no affiliation of European Health within the scope of Regulations (EEC) n° 1408/71 and 574/72 coordinating social security systems.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-07-25 (Actual); Primary Completion 2021-10-05 (Actual); Study Completion 2022-03-14 (Actual)

PRIMARY OUTCOMES:
The objective metabolic responses | at month 3
  The objective metabolic responses is the percentage of patients with a complete metabolic response, partial metabolic response (reduction of a minimum of 30% in target lesions), stable metabolic disease or progressive metabolic disease according to PERCIST criteria (Haroche, et al. 2015) at Month 3. PERCIST criteria is defined by the PET response and will be used to evaluate the overall therapeutic response at month 3.
  For PERCIST criteria, a quantitative analysis of uptake will be performed using the standard uptake value (SUV). Fitting regions of interest covering pathologic uptake will be used to define target lesions. PERCIST will be used to classify patients metabolic response.

SECONDARY OUTCOMES:
Overall survival | every 12 weeks up to 36 weeks for Cobimetinib group and 48 weeks for Placebo group
  Overall survival is defined as the time between the date of randomisation and the death.
Progression-free survival | every 12 weeks up to 36 weeks for Cobimetinib group and 48 weeks for Placebo group
  Progression-free survival is defined as the time between the date of randomisation and the first documented event of disease progression according to PERCIST criteria (Haroche, et al. 2015).
Number of participants with adverse events as assessed by CTCAE v4.0 | From the randomisation up to 36 weeks for Cobimetinib group and 48 weeks for Placebo group.
  All adverse events from clinical evaluations and laboratory measurements assessed by CTCAE v4.0
Overall response of Cobimetinib (metabolic and tumor assessment) | From the evaluation performed just before the treatment (Day 0 for Cobimetinib group, Week 12 for Placebo group)
  Overall response of Cobimetinib (metabolic and tumor assessment) assessed after 36 weeks of Cobimetinib treatment or until Cobimetinib stop.
CRP levels | At Baseline, Week 12, Week 24, Week 36 and Week 48 (for Placebo group)
  CRP levels assessed from blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Fleur Dr COHEN AUBART, Principal Investigator — APHP
Locations (1):
- Service de Médecine interne - La Pitié Salpêtrière, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jouenne F, Benattia A, Tazi A. Mitogen-activating protein kinase pathway alterations in Langerhans cell histiocytosis. Curr Opin Oncol. 2021 Mar 1;33(2):101-109. doi: 10.1097/CCO.0000000000000707. PMID 33315630